CLINICAL TRIAL: NCT03869255
Title: Nasal Carrying by Staphylococcus Aureus ST398 Strains in Community and Hospital Settings
Acronym: CONASA 398
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: API/2018/96
Record Dates: First submitted 2019-02-21; First posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-02

CONDITIONS: Staphylococcus Aureus Nasal Carriage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospitalized patients: Within 48 hours of admission to participating departments, all patiens will be included. A nasal swab will be performed within the first 48 hours and on the 7th day.
  Interventions: Procedure: Nasal swab
- Community patients: People coming to donate blood in "Etablissement Français du Sang" will be included and a nasal swab will be performed
  Interventions: Procedure: Nasal swab

INTERVENTIONS:
Procedure: Nasal swab — In hospitalized patiens, a nasal swab will be performed within the first 48 hours and on the 7th day. In community patient, only one swab will be performed

SUMMARY:
The aim of this study was to compare the prevalence of nasal carrying of SA ST398 strains in community and hospital settings, identify the factors associated with colonization of SA ST398, determine the distribution of imported and acquired cases among SA ST398 hospital cases and characterize the genetic structure of the ST398 SA population involved in colonization.

DETAILED DESCRIPTION:
Staphylococcus aureus (SA) is a ubiquitous bacterium, part of the human commensal flora. The mucosa of the anterior nasal cavities represents the preferred site of colonization of SA. The SA ST398 clone, belonging to CC 398, was initially described as a zoonotic agent initially identified in France and the Netherlands. In fact, ST398 strains are separated into two distinct populations: a methicillin-resistant SA population (SAMR) with notion of contact with animals and a more virulent methicillin-sensitive SA population (SAMS) than its counterpart, isolated from serious human infections and without notion of exposure to farm animals. Recently, we have shown that, in SA bacteremia, all strains of SA ST398 are sensitive to methicillin and that the prevalence of ST398 among all SAMS responsible for bacteremia at Besançon University Hospital increased between 2009 and 2014, increased from 4 to 15%. However, we were unable to study nasal colonization to support the mode of acquisition of SA ST398 (community vs. healthcare acquisition).

ELIGIBILITY:
For community patients :

Inclusion Criteria:

* the selection criteria for blood donation
* age ≥ 18 years old
* No refusal of the person

Exclusion Criteria:

* None

For hospitalized patients :

Inclusion Criteria:

* age ≥ 18 years old
* hospitalization in one of the services participating in the study
* no refusal of the person

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For community patients : All patients presenting for blood donation will be included For hospitalized patients, all patients hospitalized less than 48h in a service participating to the study will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients nasal carrying of SA ST398 strains in community and hospital settings | One day
  Number of patients with SA ST398 positive nasal swab in community will be compared with number of patients with SA ST398 positive nasal swab in hospital

SECONDARY OUTCOMES:
Number of patietns with specific Clinical and demographic data associated with nasal carrying of SA ST398 | One day
  Clinical and demographic (sex, age, gender, comorbidities, tabaco...) data will be compared between patients with SA ST398 positive nasal swab and SA ST398 negative nasal swab
Number of patients with SA ST398 positive nasal swab to seven days of hospitalization | 7 days
  Number of patients with SA ST398 positive nasal swab to seven days of hospitalization will be compared with the number of patients with SA ST398 positive nasal swab within the first 48 hours of hospitalization
Number of virulence gene in SA ST 398 strains | One day
  Presence of virulence gene in SA ST 398 strains

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No